CLINICAL TRIAL: NCT04237805
Title: A Phase I/II, Multi-center Clinical Study: Dose-finding Phase I Study of Foritinib Succinate in Advanced ALK-positive NSCLC Patients and Phase II Study of Foritinib Succinate in ALK or ROS1-positive NSCLC Patients
Brief Title: A Phase I/II Clinical Study of SAF-189s in Non-small Cell Lung Cancer (NSCLC) Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Fosun Pharmaceutical Industrial Development Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAF001
Record Dates: First submitted 2020-01-15; First posted 2020-01-23 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-05

CONDITIONS: Advanced Cancer; Advanced Solid Tumor; Lung Cancer, Nonsmall Cell
Keywords: ALK-rearranged; ALK-positive; ROS1-rearranged; ROS1-positive
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SAF-189s (Experimental): The phase I dose study will enrol patients with advanced malignant solid tumors that are ALK-positive, and the phase II study will be divided into two parts, Part I Some patients with ALK/ROS1 positive advanced non-small cell lung cancer were enrolled in the 210m,80mg,120mg and 160mg dose groups for safety evaluation.In the second part, two cohorts will be included and 110 ROS1 patients will be enrolled. Except for the PK induction period, all patients will receive oral administration of SAF189s once a day for a continuous period of 21 days.
  Interventions: Drug: SAF-189s

INTERVENTIONS:
Drug: SAF-189s — 20mg，40mg，80mg，120mg，160mg，210mg，once daily
  Other Names: foritinib succinate

SUMMARY:
The study comprises two phases: phase I dose escalation (including PK run-in period and treatment period) and phase II study.

DETAILED DESCRIPTION:
This is a multicenter, single-arm, open-label dose-finding phase I/II study to determine the MTD and RP2D of oral foritinib succinate monotherapy in patients with advanced ALK-positive malignant solid tumor, and to evaluate the safety, tolerability, and PK characteristics of SAF-189s in patients with advanced ALK-positive NSCLC. Phase II clinical study was conducted to evaluate the efficacy, tumor activity, and safety of remitinib succinate in patients with ALK/ROS1 positive advanced non-small cell lung cancer, and to preliminary evaluate the population pharmacokinetic characteristics of remitinib succinate.

This study consisted of two phases: phase I (including PK induction and continuous administration) and phase II, Phase I dose escalation : the patients with advanced ALK-positive malignant solid tumor who have progressed on standard therapies; Phase I study: histologically or cytologically confirmed, locally advanced ALK-positive and/or metastatic stage IIIB/IV NSCLC who have progressed on standard therapy; Phase II Study Part I: Patients with histologically and/or cytologically confirmed ALK or ROS1 positive locally-advanced and/or metastatic stage IIIb ~IV NSCLC;Patients who had not previously received or had received only one ALK/ROS1 inhibitor for disease progression or intolerance, and who had no more than 3 previous treatment lines overall Phase II Study Part Ⅱ: cohort1：ROS1-positive locally advanced and/or metastatic stage IIIB~IV NSCLC patients diagnosed histologically and/or cytologically, with no prior systemic therapy or only one line of non-ROS1-inhibitor treatment cohort 2: patients with histologically and/or cytologically confirmed ROS1-positive locally advanced and/or metastatic stage IIIb ~IV NSCLC who had previously only received crizotinib as a ROS1 inhibitor for disease progression or intolerance and had no more than 3 overall previous treatment lines；

ELIGIBILITY:
Inclusion Criteria:

1) Have a full understanding of this study and voluntarily sign an informed consent form (ICF) 2）Phase I dose escalation : the patients with advanced ALK-positive malignant solid tumor who have progressed on standard therapies; Phase I study: histologically or cytologically confirmed, locally advanced ALK-positive and/or metastatic stage IIIB/IV NSCLC who have progressed on standard therapy; Phase II Study Part I: Patients with histologically and/or cytologically confirmed ALK or ROS1 positive locally-advanced and/or metastatic stage IIIb ~IV NSCLC;Patients who had not previously received or had received only one ALK/ROS1 inhibitor for disease progression or intolerance, and who had no more than 3 previous treatment lines overall Phase II Study Part Ⅱ: cohort1：ROS1-positive locally advanced and/or metastatic stage IIIB~IV NSCLC patients diagnosed histologically and/or cytologically, with no prior systemic therapy or only one line of non-ROS1-inhibitor treatment cohort 2: patients with histologically and/or cytologically confirmed ROS1-positive locally advanced and/or metastatic stage IIIb ~IV NSCLC who had previously only received crizotinib as a ROS1 inhibitor for disease progression or intolerance and had no more than 3 overall previous treatment lines； 3) At least one measurable lesion per RECIST1.1; Note: a lesion previously treated by radiotherapy is not considered as a target lesion, unless confirmed progression is documented after radiotherapy.

4) ECOG performance score ≤ 2; 5) Male or female patients ≥ 18 and ≤ 75 years old in Phase I ；Male or female patients ≥ 18 in Phase II 6) Life expectancy ≥ 12 weeks; 7) Patient with appropriate organ function as documented by:

1. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L;
2. Hemoglobin ≥ 90 g/L;
3. Platelets (PLT) ≥ 100 × 109/L
4. Serum total bilirubin ≤ 1.5 × ULN (if the patient has Gilbert's syndrome, ≤ 3 × ULN and direct bilirubin ≤ 1.5 × ULN);
5. Aspartate aminotransferase (AST) and alanine transaminase (ALT) ≤ 2.5 × ULN (≤ 5 × ULN for patient with liver metastases);
6. Creatinine clearance (CrCL) ≥ 50 mL/min (calculated by Cockcroft-Gault equation)
7. Fasting blood glucose ≤ 200 mg/dL (≤ 11.1 mmol/L) 8) Toxicities from any prior therapy, surgery, or radiotherapy must have resolved to Grade 0 or 1 per NCI-CTCAE (Version 4.03), exception of alopecia; 9）Within 21 days prior to enrolment, women of reproductive age had to confirm a negative serological pregnancy test and agree to use an effective contraceptive method for all study drug use and for 28 days after the last dose.For the purposes of this protocol, women of childbearing age are defined as sexually mature women who: 1) have not undergone hysterectomy or bilateral oophorectomy, or 2) have natural menopause that has not lasted continuously for 24 months (amenorrhea after cancer treatment does not exclude fertility) (i.e., have had menstruation at any time during the previous consecutive 24 months);

Exclusion Criteria:

1. Has had prior chemotherapy, anti-cancer treatment with biological drugs, or other investigational agents within 28 days or received TKI or targeted therapies within 14 days prior to enrollment;
2. Received radiotherapy within 21 days prior to the 1st dose or continuance of toxicities due to prior radiotherapy that do not recover to Grade 0 or 1;
3. Patients who received major surgery within 3 weeks before enrollment or have not adequately recovered from prior surgery;
4. Patients with central nervous system (CNS) metastases requiring

   1. Clinical local intervention such as surgical excision, radiotherapy or other therapies
   2. Phase I dose escalation: patients requiring systemic treatment with corticosteroids (>10 mg/day prednisone or equivalent) are not eligible for dose escalation study (not applicable to patients participating Phase I cohort expansion or Phase II).
5. Diabetics without stable control and with insulin therapy (patients with fasting blood glucose below 7mmol/L, who are receiving stable hypoglycemic drug regimen, and whose blood glucose control is stable as evaluated by specialist doctors are allowed to be enrolled); 6）Difficulty in swallowing or having an active digestive disorder or having undergone major gastrointestinal surgery may significantly affect the administration or absorption of SAF189s (e.g. ulcerative lesions, uncontrollable nausea, vomiting, diarrhoea, malabsorption syndrome, and enteroctomies) 7）Patients who are taking the following medicines:

   1. Repaglinide (cytochrome [CYP]2C8) and drugs metabolized via CYP3A4 enzyme within 1 week before enrollment;
   2. Medicines which are known to cause QT prolongation or torsade de pointes;
   3. Coumarin anticoagulants within 1 week before enrollment (low molecular weight heparin is permitted);
   4. Illegal drugs;

8) Has a history of acute pancreatitis within 1 year before enrollment, or past history of chronic pancreatitis; 9) Patients have positive laboratory test for anti-HCV, or are diagnosed with human immunodeficiency virus (HIV) infection, or who refuse to receive HIV screen test; 10) Patients have other malignant tumor history or with other malignant tumors simultaneously; 11) Impairment of cardiac function or clinically significant heart disease, including New York College of Cardiology (NYHA) grade ≥ 3 congestive heart failure, arrhythmias, conduction abnormalities requiring treatment, cardiomyopathy, or uncontrolled hypertension； 12) Corrected QT interval using Fridericia formula > 450 msec for male patients and > 470 msec for female patients; 13) Patients have uncured interstitial lung disease history or non-infectious pneumonitis prior to enrollment, except for those induced by radiation therapy; 14）Any other clinically significant disease or condition (such as uncontrolled diabetes, active or uncontrolled infections, etc.) that the investigator believes could affect protocol adherence or affect the patient's ability to sign up for ICF; 15）Spinal cord metastases with potential risk or symptoms of spinal cord compression； 16）The second cohort received ROS1 inhibitors other than crizotinib； 17）The patient had uncontrollable amounts of pleural effusion, ascites, and pericardial effusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2016-11-14 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
DLT | 24 days after the first dose in the dose escalation phase
  Dose Limiting Toxicity incidence within 24 days after the first dose in the dose escalation phase
ORR | until 6 months' treatment of the last patients in each cohort
  Objective response rate

SECONDARY OUTCOMES:
TEAE | through study completion, an average of 3 year
  TEAE incidence, types, grade of toxicity according to NCI-CTCAE (version 5.0); study-related TEAE, SAE, study-related SAE, ≥ Grade 3 TEAE, ≥ Grade 3 TESAE, and TEAE leading to permanent discontinuation.
PFS | 3 years
  Progression-free survival (PFS)
CBR | 3 years
  clinical benefit rate (CBR)
DOR | 3 years
  duration of response (DoR)
OS | 4 years
  Overall survival (OS)
Cmax | 1 years
  Maximum Plasma Concentration
CNS responses | 4 years
  Central nervous system efficacy evaluation，（time to CNS progression，CNS TTP），（CNS objective response rate，CNS ORR）,（duration of CNS response，CNS DOR）

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, Doctor, Principal Investigator — Guangdong Province People's General Hospital
Locations (41):
- China (41):
  - he First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Guangdong Province People's General Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Cancer Hospital Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen, Guangdong
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhengzhou Central Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital/The Affiliated Cancer Hospital of Xiangya School of Medicine, Central South University, Changsha, Hunan
  - The Central Hospital of Yongzhou, Yongzhou, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - General Hospital of Xuzhou Mining Group, Xuzhou, Jiangsu
  - The second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Jilin Cancer Hospital, Jilin, Jilin
  - Yanbian University Affiliated Hospital, Yanji, Jilin
  - The first affiliated hospital of China medical university, Shenyang, Liaoning
  - Jinan Central Hospital, Jinan, Shandong
  - No. 960 Hospital of the Joint Service Support Force of Chinese People's Liberation Army, Jinan, Shandong
  - Shandong Provincial Qianfoshan Hospital, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Shanghai Chest Hospital,Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Jieyang Peoples Hospital, Jieyang, Shanxi
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - The second peoples hospital of Neijiang, Neijiang, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality
  - Tianjin Peoples Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Medical School of Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - SIR RUN RUN SHAW HOSPITAL Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Shulan (Hangzhou) Hospital, Hangzhou, Zhengjiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang JJ, Zhou J, Liu SM, Li M, Zhang Z, Cheng Y, Fan Y, Pan H, Wang B, Chen G, Wang K, Jiang L, Hu Y, Shi J, Dong X, Ding C, Liu Y, Liu Z, Liao W, Li W, Wang J, Yi S, Zhao Q, Zang A, Chen Y, Cui J, Luo P, Shen X, Sun M, Wang C, Wu YL; SAF001 study group. Foritinib in advanced ROS1-rearranged non-small-cell lung cancer in China: a multicentre, open-label, single-arm, phase 2 study. Lancet Respir Med. 2024 Sep;12(9):671-680. doi: 10.1016/S2213-2600(24)00171-1. Epub 2024 Jul 23. PMID 39059398
- [Derived] Xia ZJ, Ji YC, Sun DQ, Peng X, Gao YL, Fang YF, Zhao XD, Wang WB, Ding J, Geng MY, Ai J. SAF-189s, a potent new-generation ROS1 inhibitor, is active against crizotinib-resistant ROS1 mutant-driven tumors. Acta Pharmacol Sin. 2021 Jun;42(6):998-1004. doi: 10.1038/s41401-020-00513-3. Epub 2020 Sep 11. PMID 32918045